CLINICAL TRIAL: NCT00454714
Title: Application of Sildenafil in Patients With Documented Coronary Vasospasm to Explore the Pathophysiology of Coronary Vasospasm and the Therapeutic Effect of Sildenafil in Patients Suffering From Coronary Vasospasm
Brief Title: Therapeutic Effect of Sildenafil in Patients With Coronary Vasospasm
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study not started
Sponsor: Udo Sechtem (Other)
Responsible Party: Sponsor-Investigator, Udo Sechtem, Prof. Udo Sechtem, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Organization: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBK091
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Coronary Vasospasm
MeSH Terms: conditions — Coronary Vasospasm | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Sildenafil arm
  Interventions: Drug: single dose Sildenafil
- B (Placebo Comparator): Placebo arm
  Interventions: Drug: Single dose placebo

INTERVENTIONS:
Drug: single dose Sildenafil — Application of a single dose Sildenafil
  Arms: A
Drug: Single dose placebo — Application of a single dose placebo
  Arms: B

SUMMARY:
This will be a prospective, phase IIIb, double-blind and randomized trial testing the effect of single dose sildenafil application in patients with coronary vasospasm compared to placebo application.

The target variable to be tested is the degree of coronary vasoconstriction in response to intracoronary ACh application (in addition to clinical chest pain) which will be imaged by coronary angiography and measured using quantitative coronary angiography software.

Main objective: Has sildenafil the potency to inhibit the induction of coronary vasospasm by intracoronary ACh-application in patients with proven coronary artery spasm?

Secondary objective: Which degree of coronary vasospasm inhibition can be achieved with sildenafil?

DETAILED DESCRIPTION:
Coronary artery spasm is an abrupt severe vasoconstrictor response which may occur spontaneously in normal and diseased coronary arteries. It may result in myocardial ischemia and may be provoked by various stimuli such as acetylcholine (ACh). Coronary vasospasm is involved in the pathogenesis of Prinzmetal's angina, acute myocardial infarction or sudden cardiac death due to ventricular arrythmias and chest pain symptoms associated with viral myocarditis.

The precise cellular and molecular mechanisms of coronary vasospasm have not yet been elucidated. The most often suggested but competing explanations for this disease are coronary endothelial dysfunction secondary to impaired nitric oxide production versus coronary smooth muscle cell hyperreactivity with or without additional endothelial dysfunction. As the precise cellular mechanism is currently unknown a large group of people can currently not be treated appropriately despite the use of nitrates and calcium antagonists.

Sildenafil is a phosphodiesterase(PDE)-5 inhibitor approved for the treatment of both erectile dysfunction and pulmonary hypertension. PDE-5 has been shown to be also present and play an important vasomotor role in the coronary vessel wall. Application of the inhibitor sildenafil has been shown to increase the resting coronary artery diameter. Furthermore, atherosclerotic coronary artery segments which vasoconstrict following intracoronary ACh-application vasodilate following the application of sildenafil when ACh-testing is repeated. Other studies are also suggesting an improved endothelial function after sildenafil application for both the coronary and the peripheral vasculature.

Taken together, sildenafil is expected to have a positive effect on coronary vasomotility. Whether sildenafil can totally prevent the occurrence of coronary vasospasm or at least decrease the severity of vasospasm has not been studied so far. Thus, the aim of this study is to analyse the possible anti-spastic effects of sildenafil in patients suffering from coronary vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50y
* Framingham risk score < 10%
* no contraindication to sildenafil application
* clinical history of atypical angina pectoris
* exclusion of significant coronary artery disease (stenosis ≥ 50%) by coronary angiography
* documented coronary spasm by ACh-testing in at least one coronary artery segment
* written informed consent

Exclusion Criteria:

* existing contraindication to sildenafil application
* significant coronary artery disease (≥ 50%)
* valvular, inflammatory, dilative or other cardiomyopathies
* congestive heart failure (left ventricular ejection fraction < 60%) of any reason
* need for therapeutic treatment with nitrates or intake of any nitrates in the last 24h before coronary angiography
* participation in another clinical trial at the moment or in the last 30 days
* hypotonic blood pressure (<90/50mmHg)
* hepatic insufficiency (> Child-Pugh-classification A)
* renal insufficiency with a GFR < 60ml/min- pregnancy or lactation
* not able to consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03-01; Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of coronary vasospasm in spite of medical treatment | After inclusion of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Udo Sechtem, MD, Study Director — Robert Bosch-Krankenhaus Stuttgart
Locations (1):
- Robert-Bosch-Krankenhaus, Stuttgart, Germany